CLINICAL TRIAL: NCT05261802
Title: AVANCE-Houston FRAMEWorks Healthy Marriage and Responsible Fatherhood Program Evaluation
Brief Title: AVANCE-Houston FRAMEWorks Program Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/32
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Adults

STUDY DESIGN:
Intervention Model Description: Participants in arm 1 receive 14 hours of Survival Skills for Healthy Families curricula over 7 weeks. Participants also receive employment supports and case management services.
  Participants in arm 2 receive 14 hours of Survival Skills for Healthy Families in a compressed format during a 16-hour weekend retreat, followed by a 2-hour reflections workshop two weeks later. Participants also receive employment supports and case management services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AVANCE-Houston FRAMEWorks Program Weekly Workshop Format (Experimental): A trained facilitator, supported by Career and Family Coaches, leads every HMRE parenting workshop for adults via multiple delivery models: in recurring weekly workshops (2 hours each workshop for 7 weeks) and intensive weekend retreats (totaling 16 hours). Additionally, AVANCE offers the weekly workshops either virtually via Zoom or in-person. All workshop models were offered to program participants who were able to choose whether the weekly (either in-person or virtually) or the weekend (in-person only) format worked best for them. Curriculum content is consistent across all delivery methods and target hours for all participants is 14 hours.
  Interventions: Other: Descriptive Intervention

INTERVENTIONS:
Other: Descriptive Intervention — A trained facilitator, supported by Career and Family Coaches, leads every HMRE parenting workshop for adults via multiple delivery models: in recurring weekly workshops (2 hours each workshop for 7 weeks) and intensive weekend retreats (totaling 16 hours). Additionally, AVANCE offers the weekly workshops either virtually via Zoom or in-person. All workshop models were offered to program participants who were able to choose whether the weekly (either in-person or virtually) or the weekend (in-person only) format worked best for them. Curriculum content is consistent across all delivery methods and target hours for all participants is 14 hours.

SUMMARY:
AVANCE-Houston seeks to understand whether a standard or compressed schedule format for delivering the Survival Skills for Healthy Families curriculum better meets the needs of low-income adults to improve skill retention and, ultimately, to promote better outcomes for healthy family relationships and economic stability.

DETAILED DESCRIPTION:
AVANCE-Houston's FRAMEWorks (Family, Relationship, and Marriage Education Works) Project seeks to promote healthy family relationships and economic stability by providing the Survival Skills for Healthy Families (SSHF) curriculum to cohorts of low-income adults. Developed by Family Wellness Associates, SSHF is an evidence-based curriculum delivered through a series of workshops that focus on communication skills, conflict resolution, knowledge of the benefits of marriage, stress and anger management, parenting skills, financial literacy, job and career advancement, and relationship skills to improve family and economic stability. In the past, AVANCE has offered two curriculum delivery models: recurring weekly workshops (standard schedule format) and intensive weekend retreats (compressed schedule format). Each model meets the needs of the target population in different ways, and participants consider factors such as childcare, work/school schedules, weekend availability, and geographic location when choosing their preferred model.

The key goal of this descriptive evaluation is to assess the extent that attitudes and behaviors related to parenting, partner relationships, and financial and job readiness change after participation in the SSHF curriculum. Though the program offers support services and economic stability resources, our analysis will only include outcome changes based on surveys taken at program enrollment, program completion, and one-year post-enrollment. Additionally, a secondary analysis will focus on the ancillary question of whether differences in outcomes exist between in-person and virtual format group participants, and subgroup analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Reside in Harris County (Houston area), TX

Exclusion Criteria:

* Minor (under the age of 18)
* Reside outside of Harris County (Houston area), TX

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1682 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Parenting behavior measurement #1 | Change from baseline in parenting behavior (frequency of support for child) at 12 months from enrollment.
  How did parenting behavior outcomes change from program enrollment to 1 year after enrollment?
  Items measured include:
  Parenting behavior measured with:
  4 items - frequency of support for child (4-point scale)
  Measured on the parenting behavior scale #1 as:
  1 = Never, 2 = Hardly ever, 3 = Sometimes, 4 = Often
  The higher the rating, the better the score.
Partner relationship behavior measurement #1 | Change from baseline in partner relationship behavior (frequency of key relationship behaviors) at 12 months from enrollment.
  How did partner relationship behavior outcomes change from program enrollment to 1 year after enrollment?
  Items measured include:
  Partner relationship behavior measured with:
  3 items - frequency of key relationship behaviors (4-point scale)
  Measured on the partner relationship behavior scale #1 as:
  1 = Never, 2 = Hardly ever, 3 = Sometimes, 4 = Often
  Some items in this scale are reverse-coded. For 6 items, the higher the rating, the better the score. For 1 item, the lower the rating, the better the score.
Financial readiness measurement #1 | Change from baseline in financial readiness (presence of savings and checking accounts) at 12 months from enrollment.
  How did financial readiness behavior outcomes change from program enrollment to 1 year after enrollment?
  Items measured include:
  Financial readiness measured with:
  2 items - presence of a savings account and checking account (dichotomous)
  1 = Yes, 0 = No, so the higher the rating, the better the score.

SECONDARY OUTCOMES:
Parenting attitudes measurement #1 | Change from baseline in parenting attitudes (frequency of supportive feelings toward child) immediately after program completion.
  4A) How did parenting attitude outcomes change from program enrollment to program completion?
  Items measured include:
  Parenting attitudes measured with:
  4 items - frequency of supportive feelings toward child (4-point scale)
  Measured on the parenting attitudes scale #1 as:
  1 = Never, 2 = Hardly ever, 3 = Sometimes, 4 = Often
  The higher the rating, the better the score.
Partner relationship attitudes measurement #1 | Change from baseline in parenting attitudes (level of agreement with how supportive partner is) immediately after program completion.
  5) How did partner relationship attitude outcomes change from program enrollment to program completion?
  Items measured include:
  Partner relationship attitudes measured with:
  5 items - level of agreement with how supportive partner is (5-point scale)
  Measured on the partner relationship attitudes scale #1 as:
  1 = Strongly agree, 2 = Agree, 3 = Disagree, 4 = Strongly disagree, 5 = Not applicable
  The lower the rating, the better the score.
Job readiness behaviors #1 | Change from baseline in financial readiness (presence of savings and checking accounts) at 12 months from enrollment.
  6) How did job readiness behavior outcomes change from program enrollment to 1 year after enrollment?
  Items measured include:
  1 item - presence of a resume to give employers (dichotomous)?
  1 = Yes, 0 = No, so the higher the rating, the better the score.

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- AVANCE-Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.